CLINICAL TRIAL: NCT05546736
Title: Effects of the iCanWork Intervention to Improve Cancer Survivors' Experience With Return to Work: A Randomized Controlled Trial (RCT)
Brief Title: iCanWork: A Randomized Controlled Trial
Acronym: iCanWork
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Christine Maheu, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: iCanWork_CIHR
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Cancer-related Problem/Condition; Survivorship; Quality of Life
Keywords: return to work; cancer survivors; vocational rehabilitation; randomized controlled trial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCanWork Intervention (Experimental): iCanWork includes 6 1-hour sessions with a VRC and 1 to 4 1-hour sessions with an OT. In the positive event that a participant has returned to work during the study, three of the six VRC sessions are reserved to support the participants in their transition to the workplace.
  Interventions: Behavioral: iCanWork Intervention
- Control (No Intervention): Participants randomized to the control group will receive their usual care and will be referred to the Cancer Work website for educational resources related to RTW. If they contact the team with RTW-related questions, they will be referred to their care teams.

INTERVENTIONS:
Behavioral: iCanWork Intervention — Participants will receive RTW support from the VRC and OT.
  Arms: iCanWork Intervention

SUMMARY:
The aim of this study is to evaluate the effectiveness of the iCanWork intervention in assisting cancer survivors (CS) to return to work (RTW) and its impact on their health-related quality of life (QoL), health service utilization, RTW readiness, time to RTW, and work capacity.

DETAILED DESCRIPTION:
The iCanWork intervention comprises several elements related to health and work, taken from the latest reviews that recommend a remote and individual intervention, led by a vocational rehabilitation counsellor (VRC), experts in assisting RTW for CS. The intervention includes 6 sessions with a VRC and 1-4 sessions with an occupational therapist (OT). A total of 270 CS will be recruited into 2 groups (intervention or control). The duration of this study is 24 months. Study participants will complete electronic questionnaires measuring study variables at baseline before randomization and at 6-month, 12-month, 18-month, and 24-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with cancer (all types) treated with curative intent and of working age (between 18 and 65 at the time of diagnosis)
* gainfully employed at the time of diagnosis (full or part-time, including students)
* still on sick leave, including long-term disability leave, but for less than 2 years
* has not started to return to work, since stopping due to cancer
* can read and understand English or French
* reside in Canada.

Exclusion Criteria:

- If the cancer survivor's physicians consider returning to work unwise, such as due to a metastatic cancer diagnosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline return to work status in the course of the 24-month study | baseline, 6 months, 12 months, 18 months, 24 months
  binary variable (Yes/No)

SECONDARY OUTCOMES:
Change from baseline health related quality of life in the course of the 24-month study | baseline, 6 months, 12 months, 18 months, 24 months
  The Patient Reported Outcome Information System (PROMIS) - Preference scale is a valid, 31-item tool to measure 7 domains of quality of life (i.e., cognition, depression, fatigue, pain, physical function, sleep disturbance, and ability to participate in social roles and activities). Each of these items is measured on five levels (e.g., "never", "rarely", "sometimes", "often", "always" or "not at all", "a little bit", "somewhat", "quite a bit", and "very much"). The responses (1 to 5 on a Likert scale) were transformed into PROMIS theta scores (mean = 0 ± SD = 1) or T-Scores (mean = 50 ± SD = 10). For cognition, physical function, and ability to participate in social roles and activities, higher T-Scores (thetas) indicate more desirable outcomes. For depression, fatigue, pain, and sleep disturbance, lower T-Scores (thetas) indicate more desirable outcomes.
Change from baseline readiness to return to work in the course of the 24-month study | baseline, 6 months, 12 months, 18 months, 24 months
  The Readiness for Return-To-Work Scale is a validated 22-item measure of the readiness to return to work stages and consists of two scales; Scale A contains 13 items for individuals who are not working and Scale B includes 9 items for individuals who are working either part or full time. Each item is scored using a 5 point scale (1 = strongly disagree, 5 = strongly agree) representing a specific readiness stage: Pre-contemplation; Contemplation; Prepared for Action-Self-evaluative; and Prepared for Action-Behavioural for those not back at work and Uncertain Maintenance or Proactive Maintenance for those who are currently working. The scale provides a final score for each readiness stage by taking the mean of the items that create that factor. Higher scores associated with a readiness stage indicate higher level of beliefs associated with that stage.
Change from baseline work capacity in the course of the 24-month study | baseline, 6 months, 12 months, 18 months, 24 months
  Work capacity will be measured with the 7-item validated Work Capacity Index which measures seven domains related to the level of work capacity namely: 1) current work capacity compared to pre-cancer work capacity; 2) current work capacity compared to job demands; 3) number of physician-diagnosed health problems; 4) work disability due to illnesses; 5) days of absenteeism since stopping work due to cancer; 6) prognosis of anticipated work capacity for the next two years; and 7) psychological resources. The score of the 7 domains is summed ranging from 7 to 49 with a higher score indicating a greater capacity for work.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol will be published with an open access peer-reviewed journal
Supporting Information: Study Protocol